CLINICAL TRIAL: NCT07057193
Title: Effect of Dexmedetomidine, Ketamine or Midazolam on the Incidence and Severity of Emergence Delirium in Preschool-Aged Children Following Squint Surgeries Under Sevoflurane Anesthesia
Brief Title: Effect of Different Drugs on Emergency Delirium in Preschool Age Patient
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Asmaa Mohammed Galal El-Deen, lecturer of anesthesia and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Zagazig S
Record Dates: First submitted 2025-06-26; First posted 2025-07-09 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Emergence Delirium, Anesthesia
Keywords: emergency delirium; Dexmedetomidine; Midazolam
MeSH Terms: conditions — Emergence Delirium | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (C group) (Placebo Comparator): patients will receive 5ml of normal saline intravenous10 min before the end of the surgical procedure as placebo.
  Interventions: Other: 5ml of normal saline
- Dexmedetomidine group (D group) (Active Comparator): patients will receive intravenous dexmedetomidine (0.25 μg/kg diluted with normal saline to a volume of 5 ml solution) 10 min before the end of the surgical procedure.
  Interventions: Drug: Dexmedetomidine group (D group)
- Ketamine group (K group) (Active Comparator): patients will receive intravenous ketamine (0.25mg/kg diluted with normal saline to a volume of 5 ml solution) 10 min before the end of the surgical procedure.
  Interventions: Drug: Ketamine group (K group)
- Midazolam group (M group) (Active Comparator): patients will receive intravenous midazolam (0.05 mg/kg diluted with normal saline to a volume of 5 ml solution) 10 min before the end of the surgical procedure.
  Interventions: Drug: Midazolam group (M group)

INTERVENTIONS:
Drug: Dexmedetomidine group (D group) — patients will receive intravenous dexmedetomidine (0.25 μg/kg diluted with normal saline to a volume of 5 ml solution) 10 min before the end of the surgical procedure.
  Arms: Dexmedetomidine group (D group)
Drug: Ketamine group (K group) — patients will receive intravenous ketamine (0.25mg/kg diluted with normal saline to a volume of 5 ml solution) 10 min before the end of the surgical procedure.
  Arms: Ketamine group (K group)
Drug: Midazolam group (M group) — patients will receive intravenous midazolam (0.05 mg/kg diluted with normal saline to a volume of 5 ml solution) 10 min before the end of the surgical procedure.
  Arms: Midazolam group (M group)
Other: 5ml of normal saline — patients will receive 5ml of normal saline intravenous10 min before the end of the surgical procedure as placebo.
  Arms: Control group (C group)

SUMMARY:
Emergence delirium (ED) was first described by Eckenhoff and colleagues in the 1960s and is defined in pediatric anesthesia as 'dissociated state of consciousness in which child is irritable, uncompromising, uncooperative, incoherent, and inconsolably crying, moaning, and kicking or thrashing. The commonly reported incidence of postoperative ED in pediatric patients especially with the use of sevoflurane or desflurane was from 10% to 80% during their presence in the post-anesthesia care unit. This side effect of general anesthesia causes distressing for parents and staff and may cause parental dissatisfaction with their child's care. Children during postoperative ED have the risks of injuring themselves or their caregivers, disruption of surgical repair, operative site bleeding, removing Intravenous (iv) lines or drains and increasing pain. This behavior may require more nursing supervision, overloading nursing resources. Although postoperative ED episodes are of short duration, their prevention is essential. Children experiencing postoperative ED may exhibit new-onset maladaptive behavioral abnormalities in the postoperative period such as enuresis, night-time crying, and separation anxiety, up to 14 days post-surgery.

The risk factors to postoperative ED are patients' characters (preschool age and preexisting behavior), the surrounding environment as parental anxiety, type of anesthesia (volatile anesthetics) as sevoflurane or halothane and the type of surgery as tonsillectomy, adenoidectomy, and strabismus surgery which is one of the most commonly undertaken surgeries in pediatric patients. It may cause visual disturbance in the recovery phase, which can result. In order to diagnose ED, the presence of pain during recovery from general anesthesia must be ruled out because it leads to a change in behavior that resembles delirium. Fortunately, one of the advantages of using the Pediatric Anesthesia Emergence Delirium (PAED) scale is its ability to distinguish between the ED and the change in behavior resulting from pain, because it focuses on changes in awareness and knowledge that are not changed by pain. Prophylactic drugs against the occurrence of postoperative ED include the adjuvant use of α2 adrenoreceptor agonists such as dexmedetomidine, ketamine, midazolam, propofol, and fentanyl. The use of these drugs with them adverse effects should be weighed against the fact that postoperative ED is a self-limited disorder. Dexmedetomidine is a highly selective α2-adrenergic receptor agonist that is associated with sedative and analgesic sparing effects. It is commonly used for prevention of emergence delirium and agitation, perioperative sympatholysis, cardiovascular stabilization, and preservation of respiratory function. Ketamine is a dissociative anesthetic. Its mechanism of action is mainly via a noncompetitive antagonism of the N - methyl - D - aspartic acid (NMDA) receptor. It also targets other receptors, such as a - amino - 3 - hydroxy - 5 - methyl - 4 - isoxazolepropionic acid (AMPA) receptors, and has additional acts as an agonist of the sigma 1 receptor. It is commonly used for acute pain management, chronic pain management, prevention of ED, and postoperative nausea and vomiting. Midazolam is short acting benzodiazepine which is central nervous system depressant. It is commonly used for premedication during pediatric anesthesia, for prevention of emotional distress and ED due to its sedative and anxiolytic properties, additionally it used for reduction of the analgesic requirement and to prevent postoperative nausea and vomiting

ELIGIBILITY:
Inclusion Criteria:

* Parents or first degree relative acceptance. - Age: 3-5 years old. - Body weight: 5% -85% of BMI (kg /m2) of the same age and sex. - Sex: Both sexes. - Physical Status: Of class I and II according to American Society of Anesthesiologists (ASA) classification. - Type of surgery: Squint surgeries under sevoflurane anesthesia.

Exclusion Criteria:

* - Children with score 3 (i.e. anxious and crying) according to the three-point anxiety scale (Kain et al. 2004). - Children with preexisting abnormal behavior, psychiatric disorders, developmental delay or central nervous system diseases (epilepsy). - Children with chronic use of sedative drugs. - Children with severe respira

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 92 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
the incidence and severity of ED using the Pediatric Anesthesia Emergence Scale (PAED) Scale. | preoperative, baseline, PACU, 10, 20, 30 mins postoperative , perioperative
  the incidence and severity of ED using the Pediatric Anesthesia Emergence Scale (PAED) Scale.

SECONDARY OUTCOMES:
recovery time. postoperative pain severity | preoperative as baseline and upon arrival to PACU, then 10, 20, and 30 minutes after admission, perioperative
  Recovery time. IV. Post operative pain severity: will be assessed upon arrival to PACU, then at 10, 20, 30 min, and finally upon discharge from it. V. Hemodynamic and SpO2 changes: MAP, HR, and SpO2 will be measured the night before surgery as baseline, then intraoperative immediately before and at 5, 10, 20, 30 min after study drug administration. In the PACU, these parameters will be recorded upon arrival to PACU and then at 10, 20 min and finally upon discharge from PACU. VI. Time to discharge from PACU. VII. The degree of parents' satisfaction. VIII. The associated side effects: such as bradycardia, hypotension, peripheral blood oxygen desaturation vomiting, and allergy to the study drugs

IPD SHARING:
Plan to Share IPD: Yes
planned after the completion of the study and publication
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: planned after the completion of the study and publication
Access Criteria: principal investigator

REFERENCES:
- [Background] Yao Y, Sun Y, Lin J, Chen W, Lin Y, Zheng X. Intranasal dexmedetomidine versus oral midazolam premedication to prevent emergence delirium in children undergoing strabismus surgery: A randomised controlled trial. Eur J Anaesthesiol. 2020 Dec;37(12):1143-1149. doi: 10.1097/EJA.0000000000001270. PMID 32976205
- [Background] Wang HY, Chen TY, Li DJ, Lin PY, Su KP, Chiang MH, Carvalho AF, Stubbs B, Tu YK, Wu YC, Roerecke M, Smith L, Tseng PT, Hung KC. Association of pharmacological prophylaxis with the risk of pediatric emergence delirium after sevoflurane anesthesia: An updated network meta-analysis. J Clin Anesth. 2021 Dec;75:110488. doi: 10.1016/j.jclinane.2021.110488. Epub 2021 Sep 1. PMID 34481361
- [Background] Uakritdathikarn T, Chongsuvivatwong V, Geater AF, Vasinanukorn M, Thinchana S, Klayna S. Perioperative desaturation and risk factors in general anesthesia. J Med Assoc Thai. 2008 Jul;91(7):1020-9. PMID 18839840
- [Background] Templeton TW, Goenaga-Diaz EJ, Downard MG, McLouth CJ, Smith TE, Templeton LB, Pecorella SH, Hammon DE, O'Brien JJ, McLaughlin DH, Lawrence AE, Tennant PR, Ririe DG. Assessment of Common Criteria for Awake Extubation in Infants and Young Children. Anesthesiology. 2019 Oct;131(4):801-808. doi: 10.1097/ALN.0000000000002870. PMID 31343462
- [Background] Shukry M, Clyde MC, Kalarickal PL, Ramadhyani U. Does dexmedetomidine prevent emergence delirium in children after sevoflurane-based general anesthesia? Paediatr Anaesth. 2005 Dec;15(12):1098-104. doi: 10.1111/j.1460-9592.2005.01660.x. PMID 16324031
- [Background] Shin S, Evans F, & Mason K (2021) "Emergence delirium in pediatric patients", Anesthesia tutorial of the week; 422,. 1-6.
- [Background] Lee AC, Reduque LL, Luban NL, Ness PM, Anton B, Heitmiller ES. Transfusion-associated hyperkalemic cardiac arrest in pediatric patients receiving massive transfusion. Transfusion. 2014 Jan;54(1):244-54. doi: 10.1111/trf.12192. Epub 2013 Apr 15. PMID 23581425
- [Background] Mountain BW, Smithson L, Cramolini M, Wyatt TH, Newman M. Dexmedetomidine as a pediatric anesthetic premedication to reduce anxiety and to deter emergence delirium. AANA J. 2011 Jun;79(3):219-24. PMID 21751690
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Kim YH, Yoon SZ, Lim HJ, Yoon SM. Prophylactic use of midazolam or propofol at the end of surgery may reduce the incidence of emergence agitation after sevoflurane anaesthesia. Anaesth Intensive Care. 2011 Sep;39(5):904-8. doi: 10.1177/0310057X1103900516. PMID 21970137
- [Background] Kain ZN, Caldwell-Andrews AA, Maranets I, McClain B, Gaal D, Mayes LC, Feng R, Zhang H. Preoperative anxiety and emergence delirium and postoperative maladaptive behaviors. Anesth Analg. 2004 Dec;99(6):1648-1654. doi: 10.1213/01.ANE.0000136471.36680.97. PMID 15562048
- [Background] Fleming S, Thompson M, Stevens R, Heneghan C, Pluddemann A, Maconochie I, Tarassenko L, Mant D. Normal ranges of heart rate and respiratory rate in children from birth to 18 years of age: a systematic review of observational studies. Lancet. 2011 Mar 19;377(9770):1011-8. doi: 10.1016/S0140-6736(10)62226-X. PMID 21411136
- [Background] Fang XZ, Gao J, Ge YL, Zhou LJ, Zhang Y. Network Meta-Analysis on the Efficacy of Dexmedetomidine, Midazolam, Ketamine, Propofol, and Fentanyl for the Prevention of Sevoflurane-Related Emergence Agitation in Children. Am J Ther. 2016 Jul-Aug;23(4):e1032-42. doi: 10.1097/MJT.0000000000000321. PMID 26186683
- [Background] ECKENHOFF JE, KNEALE DH, DRIPPS RD. The incidence and etiology of postanesthetic excitment. A clinical survey. Anesthesiology. 1961 Sep-Oct;22:667-73. doi: 10.1097/00000542-196109000-00002. No abstract available. PMID 13889092
- [Background] Doerrfuss JI, Kramer S, Tafelski S, Spies CD, Wernecke KD, Nachtigall I. Frequency, predictive factors and therapy of emergence delirium: data from a large observational clinical trial in a broad spectrum of postoperative pediatric patients. Minerva Anestesiol. 2019 Jun;85(6):617-624. doi: 10.23736/S0375-9393.19.13038-6. Epub 2019 Jan 18. PMID 30665281
- [Background] Dahmani S, Stany I, Brasher C, Lejeune C, Bruneau B, Wood C, Nivoche Y, Constant I, Murat I. Pharmacological prevention of sevoflurane- and desflurane-related emergence agitation in children: a meta-analysis of published studies. Br J Anaesth. 2010 Feb;104(2):216-23. doi: 10.1093/bja/aep376. Epub 2010 Jan 3. PMID 20047899
- [Background] Bong CL, Lim E, Allen JC, Choo WL, Siow YN, Teo PB, Tan JS. A comparison of single-dose dexmedetomidine or propofol on the incidence of emergence delirium in children undergoing general anaesthesia for magnetic resonance imaging. Anaesthesia. 2015 Apr;70(4):393-9. doi: 10.1111/anae.12867. Epub 2014 Oct 14. PMID 25311146
- [Background] Aono J, Ueda W, Mamiya K, Takimoto E, Manabe M. Greater incidence of delirium during recovery from sevoflurane anesthesia in preschool boys. Anesthesiology. 1997 Dec;87(6):1298-300. doi: 10.1097/00000542-199712000-00006. PMID 9416712
- See also: Related Info — https://www.scirp.org/journal/paperinformation?paperid=100528